CLINICAL TRIAL: NCT04483726
Title: Distal Pancreatectomy, Minimally Invasive or Open, for Malignancy (DIPLOMA): a Pan-European, Randomized Controlled, Multicenter, Patient Blinded, Non-inferiority Trial
Brief Title: Distal Pancreatectomy, Minimally Invasive or Open, for Malignancy (DIPLOMA)
Acronym: DIPLOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: AIDS Malignancy Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL19_0340
Record Dates: First submitted 2020-06-23; First posted 2020-07-23 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreas; pancreatic; surgery; minimally-invasive; cancer; adenocarcinoma; laparoscopy; randomized; prospective
MeSH Terms: conditions — Neoplasms; Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIDP (Experimental): minimally invasive distal pancreatectomy
  Interventions: Procedure: minimally invasive distal pancreatectomy
- ODP (Sham Comparator): open distal pancreatectomy
  Interventions: Procedure: open distal pancreatectomy

INTERVENTIONS:
Procedure: minimally invasive distal pancreatectomy — Minimally invasive distal pancreatectomy (either laparoscopic or robot-assisted)
  Arms: MIDP
Procedure: open distal pancreatectomy — open distal pancreatectomy
  Arms: ODP

SUMMARY:
Objective: To compare MIDP with ODP regarding radical resection rate for pancreatic ductal adenocarcinoma (PDAC) in the pancreatic body or tail.

Study design: A pan-European, randomized controlled, multicenter, patient-blinded non-inferiority trial. This protocol was designed according to the SPIRIT guidelines1. Pathologists judging the primary endpoint will be blinded for the surgical approach (MIDP vs ODP). A blinded adjudication committee will assess all endpoints.

Study population: Two groups of 129 patients (258 in total) with an indication for elective distal pancreatectomy with splenectomy because of proven or highly suspected PDAC.

Intervention: Minimally invasive distal pancreatectomy (either laparoscopic or robot-assisted)

Control: Open distal pancreatectomy

DETAILED DESCRIPTION:
Rationale: Several systematic reviews have suggested superior short term outcomes after minimally invasive distal pancreatectomy (MIDP) as compared to open distal pancreatectomy (ODP) for benign and pre-malignant disease. In the literature and in a recent pan-European survey, about one third of pancreatic surgeons expressed concerns regarding the oncologic safety (i.e. radical resection, lymph node retrieval and survival) of MIDP in pancreatic cancer. Most surgeons stated that a randomized trial assessing oncologic safety in MIDP vs ODP for pancreatic cancer is needed.

Objective: To compare MIDP with ODP regarding radical resection rate for pancreatic ductal adenocarcinoma (PDAC) in the pancreatic body or tail.

Study design: A pan-European, randomized controlled, multicenter, patient-blinded non-inferiority trial. This protocol was designed according to the SPIRIT guidelines1. Pathologists judging the primary endpoint will be blinded for the surgical approach (MIDP vs ODP). A blinded adjudication committee will assess all endpoints.

Study population: Two groups of 129 patients (258 in total) with an indication for elective distal pancreatectomy with splenectomy because of proven or highly suspected PDAC.

Intervention: Minimally invasive distal pancreatectomy (either laparoscopic or robot-assisted)

Control: Open distal pancreatectomy

Main study parameters/endpoints: Primary outcome is the microscopically radical (R0, >1mm) resection rate. Main secondary outcomes are survival, lymph node retrieval, intraoperative outcomes (such as blood loss, operative time and conversion), postoperative outcomes (such as complications, time to functional recovery and hospital stay) and quality of life

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years;
* Elective indication for distal pancreatectomy for proven or suspected PDAC;
* Upfront (without induction / down-sizing radio- and/or chemotherapy) resectable PDAC in the pancreatic body or tail;
* The tumor can be radically resected via both minimally invasive or open surgery according to the local treating team;
* The patient is fit to undergo both open and minimally invasive distal pancreatectomy

Exclusion Criteria:

* score of American society of anaesthesiologists (ASA) >3;
* A medical history of chronic pancreatitis (according to the M-ANNHEIM criteria);
* Second malignancy necessitating resection during the same procedure;
* Distant metastases (M1) including involved distant lymph nodes;
* Tumor involvement or abutment of major vessels (celiac trunk*, mesenteric artery or portomesenteric vein);
* Pregnancy;
* Participation in another study with interference of study outcomes.
* Cystic lesion having undergone malignant transformation

  * the celiac trunk should be 5mm clear from tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2025-07-09 (Estimated)

PRIMARY OUTCOMES:
microscopically radical resection rate | 1 day
  R0, >1mm

SECONDARY OUTCOMES:
survival | 1 year
  Date of death
survival | 2 years
  Date of death
survival | 3 years
  Date of death
lymph node retrieval | 1 day
  Tumor positive lymph nodes retrieved
Operative time | 1 day
  Operative time from first incision to closure of the abdomen, minutes
Intraoperative blood loss | 1 day
  Intraoperative blood loss, mL (suction canister and weight of gauzes)
intraoperative outcomes | 1 day
  Total duration of the procedure, minutes
postoperative outcomes | 1 day
  Major complications
specimen size | 1 day
  Tumor size, mm
Specimen length | 1 day
  Specimen length, mm
margin | 1 day
  Distance from tumor to transection, anterior and posterior margin, mm

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Beaujon - APHP, Clichy
  - CHU Saint Eloi - Montpellier, Montpellier
  - Centre Hospitalier Orléans, Orléans
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No